CLINICAL TRIAL: NCT01221376
Title: Phase II Study for Safety and Efficacy Evaluation of Imatinib Mesylate in Children With Chronic Myeloid Leukemia (CML) Philadelphia Chromosome-positive (Ph+)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Renato Melaragno (Other)
Responsible Party: Sponsor-Investigator, Renato Melaragno, MD, Hospital Santa Marcelina
Organization: Hospital Santa Marcelina (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571ABR23T
Record Dates: First submitted 2010-10-14; First posted 2010-10-15 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Myeloid Leukemia (CML) With Philadelphia Chromosome-positive (Ph+)
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imatinib Mesylate (Experimental)
  Interventions: Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib Mesylate — Patient will receive Imatinib Mesylate, continuous-use, 260 mg/m2/day dose, maximum allowed 400 mg, for 24 months.
  Other Names: Glivec, MI

SUMMARY:
The purpose of this study is to evaluate the hematological, cytogenetic and molecular response to continuous-use of Imatinib in children with CML Ph+.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnose: suspected CML (hematology and/or myelogram and/or immunophenotyping and/or Leukocyte alkaline phosphatase [LAP]) to be confirmed, after, by cytogenetic and/or molecular biology. OBS: only CML Ph+ newly-diagnose in chronic or accelerate phase; resistant CML Ph+ to Interferon α (INF-α), Hydroxyurea and/or low-dose ARA-C in chronic or accelerate phase; CML Ph+ with cytogenetic relapse after BMT, that didn't use Imatinib previously, in chronic or accelerate phase.
2. Female patients of childbearing age, should have pregnancy test (blood βhCG) performed before treatment initiation. Effective contraception must be used. Pregnant women won't be included.
3. Karnofsky and Lansky scale: ≥40.
4. Life expectation > 8 weeks.
5. Laboratory: renal function (serum creatinine ≤ 1,5 x ULN and/or Clearance ≥70 ml/min/1,73m2), hepatic function (total bilirubin ≤ 1,5 x ULN, TGP < 3 x ULN and albumin > 2 g/dl.
6. CNS toxicity ≤ II
7. Cardiac function: normal ejection fraction.
8. Signed ICF by child legal responsible.

Exclusion Criteria:

1. Patient receiving any other tyrosine kinase inhibitor (TKI).
2. Pregnant patient or breastfeeding.
3. Patient considered incapable to follow purposed treatment.
4. Patients with molecular relapsed.
5. Medications:

   * Colony stimulating: it cannot be administered at least 1 week before treatment.
   * Anticonvulsants: Imatinib is metabolized by P-450 enzyme, thereby subject cannot receive drug that activates the P-450 system. The anticonvulsants allowed are valproic acid and benzodiazepines.
   * Anticoagulants: The use of warfarin (Marevan) is not allowed. If anticoagulant is needed, low-molecular-weight heparin (LMWH) can be used. Avoid anticoagulants with platelets < 50000.
   * INF-Α 48h before D1.
   * Hydroxyurea 24h before D1.
   * ARA-C doses >100 mg/m2 for 5-7 days, 14 days before D1.
   * Anthracyclines, Mitoxantrone or Etoposide 21 days before D1.
   * Any other chemotherapeutic agent 28 days before D1.
   * Hematopoietic Cell Transplantation (HCT) 6 weeks before D1.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the complete cytogenetic response with continuous-use of Imatinib. | Up to 12 months

SECONDARY OUTCOMES:
Evaluate the response to continuous-use of Imatinib and the toxicity and tolerability in children with CML Ph+. | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro M Arancibia, MD, Study Chair — Casa de Saúde santa Marcelina
Locations (1):
- Hospital Santa Marcelina, São Paulo, São Paulo, Brazil